CLINICAL TRIAL: NCT06800248
Title: A Phase III Single-center, Randomized, Double-Blinded, Parallel-group, Active Controlled Study to Evaluate the Efficacy and Safety of a Single Dose of Emodepside Compared to Multiple Doses of Mebendazole in Adolescent and Adult Participants With Soil-transmitted Helminthiasis
Brief Title: Efficacy and Safety of Emodepside in Participants With Soil-transmitted Helminth Infections
Acronym: TREMO-Siargao
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Bayer (Industry); Silicon Valley Community Foundation (Other); University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P2810-23B
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Trichuris Trichiura; Infection; Hookworm Infection; Ascaris Lumbricoides Infection
Keywords: Trichuris trichiura; Ascaris lumbricoides; STH; Efficacy; Safety; Hookworm; Emodepside; Soil-transmitted helminths; Roundworm; Whipworm; Mebendazole
MeSH Terms: conditions — Trichuriasis; Hookworm Infections; Ancylostomiasis; Enterobiasis | interventions — emodepside; Bay 44-4400; Mebendazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor staff, Site staff
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emodepside (Experimental)
  Interventions: Drug: emodepside (BAY 44-4400); Drug: similar placebo to mebendazole
- Mebendazole (Active Comparator)
  Interventions: Drug: Mebendazole 100 MG; Drug: matching placebo of emodepside

INTERVENTIONS:
Drug: emodepside (BAY 44-4400) — Treatment with single dose of oral 15 mg emodepside
  Arms: Emodepside
Drug: Mebendazole 100 MG — Treatment with 100 mg mebendazole orally administered b.i.d. for 3 days
  Arms: Mebendazole
Drug: similar placebo to mebendazole — Treatment with mebendazole similar placebo orally administered b.i.d. for 3 days
  Arms: Emodepside
Drug: matching placebo of emodepside — Treatment with single dose of oral emodepside matching placebo
  Arms: Mebendazole

SUMMARY:
This study aims to assess the efficacy and safety of emodepside compared to mebendazole in adults and adolescents infected with T. trichiura, either as single infection or co-infections with hookworm and/or A. lumbricoides.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant (confirmed by a negative serum pregnancy test) and non-breastfeeding female participants aged 12 years and older.
2. T. trichiura as a single infection or co-infection with hookworm and/or A. lumbricoides, confirmed by presence of T. trichiura eggs assessed by Kato-Katz thick smears from two stool samples (infection intensity defined as number of eggs per gram of stool (EPG): (1) light (1-999 EPG), (2) moderate to heavy (≥1000 EPG).
3. A minimum infection intensity of 24 eggs per gram of stool at baseline and at least two positive slides out of the four slides assessed at baseline.
4. Written informed consent signed by the participant and/or legally authorized representative(s) according to the participant's age as established per local regulations. In addition, participant's assent is required as applicable by local laws and regulations for adolescents of 12-17 years of age.
5. Women of childbearing potential must agree to use an effective, culturally appropriate contraceptive measure from at least 28 days prior to first dosage for hormonal contraceptives only and for non-hormonal contraceptive measures from screening Visit 2 until End of Study Visit.

Exclusion Criteria:

1. Presence of any systemic illnesses, renal and/or hepatic impairment, any other acute or chronic health conditions or congenital disorders which, in the opinion of the Investigator, would make the participant unsuitable for participation in a clinical study or may interfere with the efficacy, safety, and/or pharmacokinetic (PK) evaluation of the study drug.
2. Any of the following:

   1. Platelet <75,000/mm3
   2. Alanine Aminotransferase (ALT) or Serum Glutamic Pyruvic Transaminase (SGPT) >3x upper limit of normal (ULN)
   3. Total bilirubin >2xULN
   4. Estimated Glomerular Filtration Rate (eGFR) <90 ml/min/1.73 m2 (adolescents) or estimated creatinine clearance (CrCl) <90 ml/ min (adults)
3. Treatment with the following anthelminthic drugs: albendazole, mebendazole, ivermectin, within 28 days before the first dose of study intervention or planned before End of Study Visit.
4. Use of sensitive CYP3A4 substrates within 14 days before the start of the first study intervention and until at least 14 days after the last administration of study intervention.
5. Treatment with metronidazole within 2 days before the first dose of study intervention or planned before 24 hours after last administration of study intervention.
6. Previous assignment to a study intervention for another study planned to be administered during the period the participant is enrolled in this study (from date of informed consent to last follow-up).
7. Known allergy/hypersensitivity to mebendazole and/or emodepside

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cured of T. trichiura infection | Test of Cure Visit at 14 to 21 days after end of treatment
  Determined by negative Kato-Katz thick smears in two stool samples taken at the Test of Cure Visit

SECONDARY OUTCOMES:
Cured of A. lumbricoides infection | Time Frame: Test of Cure Visit at 14 to 21 days after end of treatment
  Determined by negative Kato-Katz thick smears in two stool samples taken at the Test of Cure Visit.
  This endpoint is only applicable for the subgroup of participants co-infected with A. lumbricoides at baseline.
Occurrence of TEAEs | Adverse events that occur after the first dose of study intervention up to 21 days after the last dose of study intervention
  Defined as any AE that occurred or worsened after the first dose of study intervention up to 21 days after the last dose of study intervention

OTHER OUTCOMES:
Cured of hookworm infection | Test of Cure Visit at 14 to 21 days after end of treatment
  Determined by negative Kato-Katz thick smears in two stool samples taken at the Test of Cure Visit.
  This endpoint is only applicable for the subgroup of participants co-infected with hookworm at baseline.
Egg reduction of each species of STH (T. trichiura, A. lumbricoides and hookworm infection) | Test of Cure Visit at 14 to 21 days after end of treatment
  Defined as logarithm of the number of eggs/g (+1) from stool samples taken at the Test of Cure Visit minus the logarithm of the number of eggs/g (+1) in stool samples taken at baseline. Egg reduction of A. lumbricoides and hookworm will only be calculated in participants co-infected with A. lumbricoides and hookworm at baseline, respectively.
Listing of individual plasma concentrations of emodepside | Plasma concentrations at 3, 6, 21-48 hours and 14-21 days after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, Professor, Study Director — Swiss Tropical & Public Health Institute
Locations (1):
- University of the Philippines Manila, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes
There is a data sharing agreement between Swiss TPH and PHL-IdC in place (study site). Data may be shared with other researchers upon request.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Mrimi EC, Welsche S, Ali SM, Hattendorf J, Keiser J. Emodepside for Trichuris trichiura and Hookworm Infection. N Engl J Med. 2023 May 18;388(20):1863-1875. doi: 10.1056/NEJMoa2212825. PMID 37195942
- [Background] Taylor L, Ahmada AA, Ali MS, Ali SM, Hattendorf J, Mohammed IS, Keiser J. Efficacy and safety of emodepside compared with albendazole in adolescents and adults with hookworm infection in Pemba Island, Tanzania: a double-blind, superiority, phase 2b, randomised controlled trial. Lancet. 2024 Aug 17;404(10453):683-691. doi: 10.1016/S0140-6736(24)01403-X. PMID 39153818